CLINICAL TRIAL: NCT05985291
Title: BurstDRTM Spinal Cord Dorsal Column Stimulation for Painful Diabetic Neuropathy
Brief Title: BurstDR Stimulation for Painful Diabetic Neuropathy
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left Advocate Health
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00104842; 23-817 (Other: Aurora IRB)
Record Dates: First submitted 2023-07-06; First posted 2023-08-14 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Painful Diabetic Neuropathy
Keywords: neurostimulation; spinal cord stimulation; burst stimulation
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Carubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PDN treated with SCS and CMM: Painful diabetic neuropathy patients treated with burst stimulation along with conservative medical management as part of regular medical care.
  Interventions: Combination Product: SCS in combination with CMM

INTERVENTIONS:
Combination Product: SCS in combination with CMM — Subjects receiving BurstDR spinal cord dorsal column stimulation in combination with conservative medical management for the treatment of painful diabetic neuropathy as part of regular medical care.

SUMMARY:
This study aims to demonstrate treatment outcomes of Painful Diabetic Neuropathy (PDN) patients treated with BurstDRTM Spinal Cord Dorsal Column Stimulator (SCS) along with conservative medical management per standard of care.

DETAILED DESCRIPTION:
In this study, we aim to systematically collect real world, observational and prospective data on the safety and effectiveness of an SCS system for the management of PDN. This study will provide, to the best of our knowledge, the first clinical, real world, prospective data in treatment of PDN with an SCS system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lower extremity Painful Diabetic Neuropathy (PDN) with symptoms for at least a year prior to signing the consent form
* PDN refractory to FDA approved medications: duloxetine, pregabalin, tapentadol, and capscaicin
* Lower limb pain intensity of 5 cm or more on a 10-cm visual analogue scale (VAS)
* HbA1c ≤10%
* BMI <45 kg/m2
* Be 22 years of age or older at the time of enrollment
* Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
* Be capable of subjective evaluation, able to read and understand English-written questionnaires, and able to read, understand and sign the written informed consent in English
* Be willing and capable of giving informed consent
* Be willing and able to comply with study-related requirements, procedures, and scheduled visits
* Have adequate cognitive ability to use a patient programmer and recharger as determined by the Investigator
* Be on a stable analgesic regimen, as determined by the Investigator, for at least 30 days prior to assessing pain intensity, and be willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device
* Have stable neurological status measured by motor, sensory and reflex function as determined by the investigator

Exclusion Criteria:

* Current daily opioid dosage greater than 120 mg morphine equivalents
* Have an average pain intensity of ≥ 3 out of 10 cm on the VAS in the upper extremities due to diabetic neuropathy at enrollment
* Have a diagnosis of a lower limb mononeuropathy (e.g., causalgia and tibial or peroneal neuropathies), have had a lower limb amputation other than toes due to diabetes, or have large (≥3 cm) and/or gangrenous ulcers of the lower limbs.
* Have a current diagnosis of a progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, central deafferentation syndrome, Complex Regional Pain Syndrome, acute herniating disc, severe spinal stenosis and brachial plexus injury, as determined by the Investigator
* Have a current diagnosis or condition such as a coagulation disorder, bleeding diathesis, platelet dysfunction, low platelet count, severely diminished functional capacity due to underlying cardiac/pulmonary disease, symptomatic uncontrolled hypertension, progressive peripheral vascular disease or uncontrolled diabetes mellitus that presents excess risk for performing the procedure, as determined clinically by the Investigator
* Be benefitting from an interventional procedure and/or surgery to treat lower limb pain (Subjects should be enrolled at least 30 days from last benefit).
* Have an existing intrathecal pain pump and/or another active implantable device such as a pacemaker
* Have a condition currently requiring or likely to require the use of diathermy or MRI that is inconsistent with ProclaimTM system guidelines in the Physician's Manual
* Have either a metastatic malignant neoplasm or untreated local malignant neoplasm
* Have a life expectancy of less than one year
* Have within 6 months of enrollment a significant untreated addiction to dependency producing medications, alcohol or illicit drugs
* Be concomitantly participating in another clinical study
* Be involved in an injury claim under current litigation
* Be a recipient of temporary Social Security Disability Insurance (SSDI) benefits due to chronic pain
* Have a pending or approved worker's compensation claim
* Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome, as determined by a psychologist in the last 12 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients older than 21 suffering from Painful Diabetic Neuropathy.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Average change from baseline to 3 months in treatment responder rates | 3 months
  Responder is defined as a subject who has at least 50% reduction in lower limb pain from baseline as measured by a 10 cm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Average change from baseline to 6 months in treatment responder rates assessed by Visual Analog Scale (0-10 cm) | 6 months
  0 no pain at all, 10 worse pain imaginable

OTHER OUTCOMES:
Percentage of patients with change from baseline in sensory neurological assessment at 3 months | 3 months
  Assessed by the healthcare provider.
Average change from baseline to 3 months in severity of neuropathic pain as measured by Neuropathic Pain 4 Questions (DN4) (0-10) | 3 months
  score of 4 or greater indicates neuropathic pain
Average change from baseline in CGM metrics from AGP report at 3 months | 3 months
Average change from baseline in health-related quality of life at 3 months as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 3 months
Average change in proportion of remitters (remission is defined as having a lower limb pain Visual Analog Score score ≤ 2.5 cm) at 6 months | 6 months
Average change in health-related quality of life as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS-29) at 6 months | 6 months
Average change from baseline to 3 months in opioid dosage measured in total morphine milligram equivalents (MME) | 3 months
Proportion of participants with clinically meaningful improvement on sensory neurological examination as determined by the investigator at 6 months compared to baseline. | 6 months
Average change from baseline to 6 months in opioid dosage measured in total MME | 6 months
Average change from baseline to 6 months in severity of neuropathic pain as measured by DN4 | 6 months
Difference in average percentage change from baseline in CGM metrics from AGP report at 6 months | 6 months
Assessment of subject outcomes satisfaction as measured through Patient Global Impression of Change (PGIC) (1-7 where higher scores mean better outcome) at 3 months and 6 months. | 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Aman, MD, Principal Investigator — Aurora Healthcare
Locations (1):
- Aurora Health Oshkosh, Oshkosh, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided